CLINICAL TRIAL: NCT04345003
Title: MR Elastography Parameters Impact on MR-HIFU Efficacy in Uterine Fibroids
Acronym: ELASTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2018/35
Record Dates: First submitted 2020-03-16; First posted 2020-04-14 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Uterine Fibroid
Keywords: HIFU; Fibroid treatment; MR elastography; Perfusion; Diffusion weighted imaging; ARFI; Fibroid stiffness
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myoma elastography (Experimental): The standard pre-therapeutic assessment includes a pelvic US to eliminate the presence of calcification of fibroids. If this absence is confirmed, the elasticity of uterine myoma (by ARFI method) will be measured.
  The standard pre-therapeutic MRI performed allows to classify and measure the myoma in order to determine if it is accessible for HIFU treatment. MRI elastography sequence with the Resoundant® system will be performed during this exam.
  Interventions: Device: Myoma elastography

INTERVENTIONS:
Device: Myoma elastography — The standard pre-therapeutic assessment includes a pelvic US to eliminate the presence of calcification of fibroids. If this absence is confirmed, the elasticity of uterine myoma (by ARFI method) will be measured.
  The standard pre-therapeutic MRI performed allows to classify and measure the myoma in order to determine if it is accessible for HIFU treatment. MRI elastography sequence with the Resoundant® system will be performed during this exam.

SUMMARY:
Magnetic resonance (MR)-guided high-intensity focused ultrasound (HIFU) ablation for fibroids is an outpatient approach for controlling symptom with an excellent safety record. It is important to exclude in advance patients who would not benefit from this treatment. For that purpose this study assesses the influence of fibroid elasticity and diffusion on ablation efficiency during treatment by MR-HIFU

DETAILED DESCRIPTION:
Pre-procedural predictors of treatment efficacy will be useful for excluding in advance patients who would not get benefit of this treatment. It seems that elastography, cellular density and perfusion could be considered as predictors. Fibroid elastography will be quantified by MRE Resoundant® system and pelvic ultrasound. Perfusion and cellular density will be quantified by MR diffusion.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Aged more than 18 years
* Not postmenopausal
* Having one or two symptomatic fibroid with size < 15cm.
* Leiomyoma type Funaki 1 or 2 on pre-therapeutic MRI
* Normal cervicovaginal smear performed within 2 years prior to inclusion
* Myoma technically accessible to MR-HIFU treatment verified on pre-therapeutic MRI
* SSS score on UFS-Qol ≥ 10
* Signed informed consent prior to any study related procedure
* With a medical insurance

Exclusion Criteria:

* Contraindicated to MR examination, gadolinium contrast injection (pregnancy etc..).
* Presence or suspicious of pelvic malignant tumor
* Myomas causing haemorrhage (meno-metrorrhagia) associated with anemia (Hb <10g/dl)
* Pregnant or lactating woman
* Small submucous myoma accessible for hysteroscopic treatment.
* Active pelvic infection
* Presence of calcification, surgical staples, or rigid implant in the passage of the ultrasound beamo People placed under legal protection, or participating in another research protocol including an exclusion period still in progress at pre-inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Composite criteria | Baseline
  Composite criteria measured from:
  * myoma stiffness (measured by Resoundant system) and
  * ablathermy efficiency.

SECONDARY OUTCOMES:
leiomyoma stiffness measured by Resoundant system | Baseline
  leiomyoma stiffness measured by Resoundant system
leiomyoma stiffness measured by ARFI-US | Baseline
  leiomyoma stiffness measured by ARFI-US
clinical efficiency | month 6
  Defined as a decrease of 10pts on UFS-Qol score
inter-observer reproducibility | Baseline
  inter-observer reproducibility of leiomyoma stiffness measurements by Resoundant system
leiomyoma perfusion | Month 6
  leiomyoma perfusion (diffusion)
leiomyoma T2 signal | Month 6
  It will be evaluated in two ways:
  The first consists of a qualitative analysis taking as a reference the signal of the paravertebral muscles. Myomas will then be classified into a hypersignal, iso-signal or hyposignal group as compared to muscles (qualitative method according to the classification of Funaki).
  The second will be a quantitative method. One ROI will be positioned in the myoma and a second in the paravertebral muscle and the ratio of these values will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No